CLINICAL TRIAL: NCT05637528
Title: Evaluating the Use of Magnetic Resonance Imaging and Contrast Enhanced Mammography After MagTrace® Use
Acronym: MagTrace2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Yvonne Vissers, Principal investigator, Zuyderland Medisch Centrum
Other Study IDs: NL82061.096.22
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Magtrace; MRI; Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MagTrace patients: Patients who underwent sentinel lymph node biopsy with MagTrace one year ago.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Patients will undergo an MRI and mammography one year after MagTrace injections
  Other Names: Mammography

SUMMARY:
Rationale: MagTrace® will be implemented as standard of care for sentinel lymph node biopsy, since it has several advantages compared to a radioactive technique. However, MagTrace® is known to interfere with MRI during follow-up imaging when using 2 mL. No data is available for patients who received 1 mL of MagTrace®, as is described in our current protocol. A contrast enhanced mammography (CEM) could be an alternative for MRI if it still shows artefacts.

Objective: The primary objective in this trial is to evaluate the use of MRI and contrast enhanced mammography after using MagTrace® to perform a sentinel node biopsy.

Study design: Prospective trial in an outpatient clinic setting.

Study population: Patients who were included in the previous MagTrace study will be asked to participate in this subsequent trial.

Study procedure: Participants will undergo MRI and CEM as standard 1-year follow-up. Since the MagTrace study started in August 2021 and finished in February 2022, this trial will start August 2022 to February 2023.

Main study parameters/endpoints: To evaluate the use of MRI and CEM, the following primary endpoints will be assessed: Visibility and size of artefacts undergoing MRI and CEM and its consequences of the quality for image assessment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Since MagTrace® will be implemented as standard localisation technique for breast conserving surgery and sentinel lymph node biopsy in Zuyderland MC, the information obtained from this trial is essential for the follow-up planning of all breast cancer patients. Therefore, the burden for the patients (undergoing extra imaging) will be in proportion to the added value of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Female patients of 18 years and older.
* Previously underwent sentinel lymph node biopsy using MagTrace®.
* Undergoing standard follow-up for previous breast cancer

Exclusion Criteria:

* Unable to comprehend the extend and implications of the study and sign for informed consent.
* Standard MRI exclusion criteria:

  * Implantable (electrical) devices (e.g., pacemaker, cochlear implants, neurostimulator);
  * Any other metal implants;
  * Claustrophobia;
  * MR-incompatible prosthetic heart valves.
* Standard CEM exclusion criteria:

  * Breast implants.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the previous MagTrace study will be included. All patients will be approached before their 1-year follow-up appointment at the radiology department. Patients will be informed by telephone by the coordinating investigator. If they are interested in this study, the patients will receive the patient information folder. Forty patients were included in the MagTrace study, so depending on the participants' willingness to participate in this subsequent trial, up to 40 patients will participate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-11-23 (Estimated); Primary Completion 2023-02-23 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Are there any artefacts visible when undergoing an MRI? | One year after surgery
  Visible artefacts on MRI
Are there any artefacts visible when undergoing a CEM? | One year after surgery
  Visible artefacts on CEM

SECONDARY OUTCOMES:
Size of the possible artefact. | One year after surgery
  Size of the artefacts on MRI and mammography
The possibility to assess the imaging by a trained radiologist | One year after surgery
  The radiologist will score the assessability using a 4 point scoring system:
  0. No artefact
  1. Good diagnostic quality
  2. Impaired but still readable
  3. Hampered clinical assessment

IPD SHARING:
Plan to Share IPD: No